CLINICAL TRIAL: NCT03700398
Title: Early Detection of Oropharyngeal and Hypopharyngeal Superficial Squamous Cell Carcinoma in Patients With Esophagus Squamous Cell Carcinoma by White Light Imaging and Optical Enhancement(OE)
Brief Title: Early Detection of Head and Neck Superficial Squamous Cell Carcinoma in Patients With Esophagus Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017SDU-QILU-06
Record Dates: First submitted 2018-09-23; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Optical Enhancement Endoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first OE (Experimental)
  Interventions: Device: first OE
- First WLI (Other)
  Interventions: Device: first WLI

INTERVENTIONS:
Device: first OE — optical enhancement(OE)，a kind of electron straining endoscopy
  Arms: first OE
Device: first WLI — the routine in the clinical practice
  Arms: First WLI

SUMMARY:
the investigators randomly divide the eligible objects into two groups:1. objects in this group will first receive OE endoscopy observation and subsequent white light imaging(WLI) observation during oropharynx and hypopharynx; 2. objects in this group will first receive WLI observation and subsequent OE observation during oropharynx and hypopharynx. Then, the investigators will compare the detect rate of oropharyngeal and hypopharyngeal superficial squamous cell carcinoma of two groups to find if OE endoscopy can improve the detect rate of oropharyngeal and hypopharyngeal superficial squamous cell carcinoma in esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* order than 18 years old
* Previous or current histopathological pathology confirmed the presence of esophageal squamous cell carcinoma

Exclusion Criteria:

* Previously confirmed pharynx/oropharyngeal squamous cell carcinoma
* Advanced pharynx/hypopharyngeal squamous cell carcinoma
* Pregnant women and lactating women
* pharyngeal or esophageal stenosis, esophageal varices, or active digestive tract hemorrhage influence the observation or fail to obtain pathological diagnosis
* Previous chemotherapy or radiation therapy affected observation
* Not completed gastroscopy or refused to take biopsy for various reasons
* Mental illnesses such as anxiety and depression affect the endoscopic observation
* Severe systemic disease, can not tolerate gastroscopy
* Refusal to sign informed consent books

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
detect rate | 12 months
  the detect rate of oropharyngeal and hypopharyngeal superficial squamous cell carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China